CLINICAL TRIAL: NCT04058106
Title: The Effect of Propofol Based Total Intravenous Anesthesia for Neuromonitoring on the Intraoperative Water Homeostasis in in Spine Surgery
Brief Title: Water Homeostasis in Propofol Based Total Intravenous Anesthesia
Status: Withdrawn | Type: Observational
Why Stopped: NO Participants Enrolled
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Myoung Hwa Kim, Department of Anesthesiology and Pain Medicine, Gangnam Severance Hospital
Other Study IDs: 3-2019-0142
Record Dates: First submitted 2019-07-23; First posted 2019-08-15 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Spine Surgery With Neuromonitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A patient who need the spine surgery: A patient who go the propofol based total intravenous anesthesia due to intraoperative neuromonitorung for spine surgery
  Interventions: Procedure: A patient who need the cerebral artery aneurysm clipping surgery

INTERVENTIONS:
Procedure: A patient who need the cerebral artery aneurysm clipping surgery — A patient who go the propofol based total intravenous anesthesia due to intraoperative neuromonitorung for unruptured cerebral artery aneurysm clipping surgery

SUMMARY:
Previous study reported that propofol binded to glutamate receptors in the hypothalamus and inhibits AVP release mediated by endogenous γ-aminobutyric acid, as well as directly inhibits the regulated calcium currents leading to normal neuronal depolarization and AVP release. However, there is no clinical data demonstrating the mechanism of propofol can induce transient DI by inhibiting the release of AVP from the hypothalamus when applied to humans. Remifentanil, binding to the μ-receptor or partly κ-receptor, have been used in total intravenous anesthesia combined with propofol, also reported inhibiting AVP relaese in both the hypothalamus (κ receptor mediator mechanism) and posterior pituitary (μ receptor mediator mechanism). However, the effects of anesthetics on water homeostasis during surgery have been not well established. Therefore, we aim to investigate the changes of intraoperative water homeostasis, and related hormones and osmolality in patients with propofol based total intravenous anesthesia due to neuromonitoring for spine surgery.

DETAILED DESCRIPTION:
"All patients will get the total intravenous anesthesia with propofol-remifentanil via an effective site-controlled infusion (TCI). For this, TCI continuous infusion pump will be used with Schnider pharmacokinetic model for propofol and Minto pharmacokinetic model for remifentanil. Propofol and remifentanil will be initiated with target effective site concentrations of 3 μg.ml-1 and 3 ng.ml-1, respectively, and controll these concentrations considering patient's consciousness loss and vital signs. And then 0.6 mg kg-1 rocuronium for muscle relaxation will be administered for intubation. Anesthesia will be maintained with BIS level 40-60 and vital signs will not be more than 20% of the baseline or less. In order to prevent the sudden movement of the patient during surgery, rocuronium will be infused continuously about 50% of TOF until the end of intraoperative neuromonitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients, ASA Classification I-Ⅲ between 20 and 70 years, scheduled the neuromonitoring for spine surgery in department of neurosurgery

Exclusion Criteria:

Taking thiazide/ACEi /ARB for hypertension

* Receiving insulin treatment due to diabetes mellitus
* Diagnosed with kidney disease or GFR < 60
* Diagnosed with liver disease or AST/ALT > 100
* Receiving furosemide or mannitol before surgery
* DI was diagnosed before surgery or having polyuria
* Taking lithium or antibiotics that are known to cause DI
* Do not understand Korean language
* Vulnerable subjects who are unable to obtain consent forms

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who undergo spine surgery with neuromonitoring
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
The water homeostasis changes of patients during propofol based total intravenous anesthesia for neuromonitoring in spine surgery | The change over time during surgery: baseline (before operation, T1), one hour after operation (T2), two hours after operation (T3), and three hours after operation (T4) - measure at four times
  The amount of urine (polyuria standard> 5 ml/kg/h) during surgery

SECONDARY OUTCOMES:
Postoperative polyuria (or diabetes insipidus) | At postoperative 24 hours and 48 hours
  Incidence of postoperative polyuria (or diabetes insipidus)

CONTACTS AND LOCATIONS:
Locations (1):
- Myoung Hwa Kim, Seoul, South Korea